CLINICAL TRIAL: NCT01781481
Title: The Pediatric Intermed: A New Clinical Decision Making Tool for Proactive Evaluation of Psychosocial Stress in Children With Inflammatory Bowel Disease
Brief Title: The Pediatric Intermed: A New Clinical Decision Making Tool
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Principal Investigator, Janice S.Cohen, Psychologist, Children's Hospital of Eastern Ontario
Other Study IDs: 09/32E
Record Dates: First submitted 2013-01-23; First posted 2013-02-01 (Estimated); Results first posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Inflammatory Bowel Disease
Keywords: Psychosocial Stress and Adjustment; Pediatric Chronic Illness; Decision-support tool; Integrated Health Care; Case Complexity
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children and youth with IBD: Children/youth (ages 8-17) with confirmed diagnoses of IBD.

SUMMARY:
The investigators have recently developed a paediatric adaptation of the INTERMED tool to address the unique developmental and social contexts of children and youth. The Pediatric INTERMED adopts a life-chart methodology to structure and organize complex case material in time, colour-coding domains to facilitate identification of areas of high need and risk for each patient. The focus of the present study is to examine the characteristics and usefulness of the tool in identifying psychosocial stress in children/youth diagnosed with Inflammatory Bowel Disease (IBD), as well as identifying overall case complexity. Children and parents will participate in a semi-structured structured interview with a clinical nurse who will then rate the 34-PIM items. To examine the construct validity of each of the Pediatric INTERMED domains (biological, psychological, social, caregiver/family, health care system) participants will complete questionnaires assessing social and psychological functioning, parent and family stress, quality of life and adaptive functioning. Information about disease status, and health care utilization will be obtained from medical chart review. It is hypothesized that greater case complexity will be predictive of more complex disease course/treatment, poorer quality of life, and increased health care utilization.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (Crohn's disease/ulcerative colitis) manifests itself in children and adolescents in up to 1/3 of those that will eventually develop these conditions. It is fast becoming an increasing problem with a 50% increase in Crohn's disease diagnosed in young children in the last decade. The patient's chronic symptoms can be both due to and result in increased child and family psychosocial stress. Similarly, treatments may add to psychosocial stress. Failure to address these psychosocial issues can lead to greater risk for poor treatment adherence, higher utilization of health care, and increased psychiatric co-morbidity. As such, improvement in health care providers' capacity to identify factors contributing to case complexity offers significant potential for improving outcomes.

Assessment of biological, psychological, social and health delivery of children's chronic illness has not been consistently integrated into the health care system. Physical and mental health services are often disconnected. Identifying those who would benefit from a mental health referral typically rests on the primary care physician or specialist and is often triggered by crises. There is also variability in physician education and comfort level in assessing psychosocial issues and especially in children with chronic illnesses in which symptoms of physical disease and mental health can overlap. Oftentimes this leaves the most responsible physician wanting for a simple assessment tool to try and determine who might be at risk and benefit from mental health intervention.

The adult INTERMED is a clinical decision-support tool that provides indicators of biological, psychological, social, heath care needs, as well as an overall index of case complexity. The tool is efficient to administer and has been successfully used by varied health care professionals in diverse medical settings to detect psychosocial needs, facilitate referral to effective services and improve health practices and outcomes. However, there is no comparable validated tool for use with children/youth.

The investigators have recently developed a pediatric adaptation of the adult INTERMED to address the unique developmental and social contexts of children and youth. A Delphi group of international experts in the field of pediatric chronic illness has reviewed the instrument to ensure clinical relevance, utility and communication clarity. Initial pilot data has demonstrated the Pediatric INTERMED has very good item inter-rater reliability. The focus of the current study is to examine the usefulness of this tool to identify biopsychosocial needs in IBD children/youth. Canada has a very high IBD incidence and prevalence. Given the facts that children with IBD face an unpredictable disease course, complex symptoms and difficult management regimens that can significantly impact their lives, it is not surprising that patients with this chronic incurable condition are highly vulnerable to mental health comorbidities. The development of this new tool will have significant importance if it proves to be useful in this population. The current study will examine a sizeable cohort of patients with regards to the relations between Pediatric INTERMED domains and other measures of children's disease, mood, behaviour, quality of life, family stress and strengths, and health services utilization. Both ulcerative colitis and Crohn's disease in children and youth lend themselves very well to this study because of the validated measures of disease severity that have been developed already.

Implementation of the novel Pediatric INTERMED n clinical practice will provide a new way to assist IBD Teams in screening their patients to be proactive in referral to mental health resources, and facilitate case management which targets patient needs. Clearly, clinicians are well aware that compliance, anxiety and depression will affect disease outcomes and too often these are only dealt with at times of crisis that has led to disease flare or reports that medicines are no longer effective. Use of this structured assessment tool begins to realize the potential of developing a truly integrated biopsychosocial approach to this chronic disease. The ease of use and objective nature of the tool will enhance communication among primary and tertiary providers and contribute to best practice approaches in the provision of integrated physical and mental health care. It will also assist in monitoring the impact of childhood chronic illness, identify factors linked to optimal health outcomes and inform program planning and resource allocations.

Study Design

Children/youth (ages of 8-17) followed in the IBD Clinic at the Children's Hospital of Eastern Ontario (CHEO) with confirmed diagnoses of IBD (Crohn's disease or ulcerative colitis) are eligible for the study. A clinical nurse will complete the Pediatric INTERMED for all study participants: based on information obtained from a review of the patients' hospital chart and a semi-structured interview conducted with the child/youth and primary caregivers), Following the Pediatric INTERMED interview, children/youth and parents participating in the project will complete a battery of self-report instruments to provide assessments of patients' social and psychological functioning, parent/family stresses, adjustment and resources. In addition, information will be obtained from the patients' charts about aspects of their diagnoses, treatment regimens, disease activity and complications, and health care utilization in the 3 months prior to their participation in the study.

Primary Hypotheses/Objectives and Statistical Rationale

1. Demonstrate that the Pediatric INTERMED is a reliable tool for use in IBD children (good inter-rater reliability and internal consistency). 40 interviews with the clinical research nurse will be videotaped so that a second health care professional trained in the use of the PIM, can also complete the PIM tool, in order to examine inter-rater reliability. Agreement between raters will be measured by means of intraclass correlations. Items within each domain will be examined to confirm that they meet internal consistency criteria (Cronbach's Alpha of .80).
2. Demonstrate that the Pediatric INTERMED domains successfully identify patient needs. Concurrent validity of the Pediatric INTERMED will be examined by looking at the Spearman rank, Pearson correlations, as appropriate, between each domain score and the measures hypothesized to be conceptually linked to the domain. To assess aspects of the Psychological Domain, the patients will complete the Children's Depression Inventory, the Multidimensional Anxiety Scale for Children and parents will complete the Child Behaviour Checklist (CBCL). Measures linked to the Social Domain of the PIM, include The Functional Disability Inventory, which taps the child's involvement in daily activities, and CBCL Competence Scores (Social, School, Activities), and the IMPACT-III, an IBD specific quality of life measure. To examine constructs linked to the Caregiver/Family Domain parents will complete the Pediatric Inventory for Parents, an index of childhood illness-related parenting stress, the Family Inventory of Life Events and Changes and the Family Inventory of Resources for Management. Disease/treatment and health care data gathered will be used to validate the Biological and Health System Domains.
3. Demonstrate that Pediatric INTERMED Complexity score is predictive of increased health care utilization. A general linear approach will be used to study the relation of the Pediatric INTERMED to health service utilization. Multivariate models will also be tested including potential covariates such as disease severity, time since diagnosis.

Statistical Power Calculations

The CHEO GI clinic sees 40 to 60 new patients diagnosed with IBD per year. In 2007 the clinic actively followed 265 children with IBD. Once diagnosed children are followed on an ongoing basis. The frequency of follow-up appointments varies depending on the nature and course of a child's disease, but the children/youth are seen at minimum three times each year. In general, participation rates in studies of children/youth with chronic illness are typically in the vicinity of 80-90% or better and this figure is consistent with the experience of the CHEO IBD clinic in the recruitment of patients into various knowledge generation studies. The PIM involves 5 domains of information inclusive of various components. To achieve significance with the various domains the investigators estimated that a total of 140-150 children will need to be enrolled. This sample size is sufficient to ensure that there are a sufficient number of observations per variable to conduct multivariate analyses. Tabachnick and Fidell (2007) and others indicated that 4 is the absolute minimum number of observations per variable to conduct multivariate analyses. A subject size of 140-150 would be sufficient to provide 4 observations per variable. Further, the anticipated sample size is sufficient to conduct all proposed analyses. Further corrections for multiple testing will be applied on a per-analysis basis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of IBD (Crohn's or Ulcerative Colitis)
* fluency in English or French
* between the ages of 8 and 17
* residing in the CHEO catchment area.

Exclusion Criteria:

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children between the ages of 8 and 17 who are followed in the CHEO GI Clinic and who have been diagnosed with an Inflammatory Bowel Disease (Crohn's Disease or Ulcerative Colitus). Once diagnosed, children are followed on an ongoing basis in the clinic for management of their chronic illness, with the frequency of follow-up appointments varying depending on the nature and course of a child's disease. Both parents of the subjects will be invited to participate in the study, although if only one parent is present only they will be included. If a child/youth is in foster placement, consent will be obtained from child protection officials to have the caregiver (s) most involved with the child/youth participate in the interview.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2010-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice S Cohen, Ph.D., Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szigethy E, Craig AE, Iobst EA, Grand RJ, Keljo D, DeMaso D, Noll R. Profile of depression in adolescents with inflammatory bowel disease: implications for treatment. Inflamm Bowel Dis. 2009 Jan;15(1):69-74. doi: 10.1002/ibd.20693. PMID 18831071
- [Background] Benchimol EI, Guttmann A, Griffiths AM, Rabeneck L, Mack DR, Brill H, Howard J, Guan J, To T. Increasing incidence of paediatric inflammatory bowel disease in Ontario, Canada: evidence from health administrative data. Gut. 2009 Nov;58(11):1490-7. doi: 10.1136/gut.2009.188383. Epub 2009 Aug 2. PMID 19651626
- [Background] Astin JA, Soeken K, Sierpina VS, Clarridge BR. Barriers to the integration of psychosocial factors in medicine: results of a national survey of physicians. J Am Board Fam Med. 2006 Nov-Dec;19(6):557-65. doi: 10.3122/jabfm.19.6.557. PMID 17090789
- [Background] Fischer CJ, Stiefel FC, De Jonge P, Guex P, Troendle A, Bulliard C, Huyse FJ, Gaillard R, Ruiz J. Case complexity and clinical outcome in diabetes mellitus. A prospective study using the INTERMED. Diabetes Metab. 2000 Sep;26(4):295-302. PMID 11011222
- [Background] Stiefel FC, Huyse FJ, Sollner W, Slaets JP, Lyons JS, Latour CH, van der Wal N, de Jonge P. Operationalizing integrated care on a clinical level: the INTERMED project. Med Clin North Am. 2006 Jul;90(4):713-58. doi: 10.1016/j.mcna.2006.05.006. PMID 16843771
- [Background] Stiefel F, Zdrojewski C, Bel Hadj F, Boffa D, Dorogi Y, So A, Ruiz J, de Jonge P. Effects of a multifaceted psychiatric intervention targeted for the complex medically ill: a randomized controlled trial. Psychother Psychosom. 2008;77(4):247-56. doi: 10.1159/000129658. Epub 2008 Apr 28. PMID 18443391
- [Background] Turner D, Otley AR, Mack D, Hyams J, de Bruijne J, Uusoue K, Walters TD, Zachos M, Mamula P, Beaton DE, Steinhart AH, Griffiths AM. Development, validation, and evaluation of a pediatric ulcerative colitis activity index: a prospective multicenter study. Gastroenterology. 2007 Aug;133(2):423-32. doi: 10.1053/j.gastro.2007.05.029. Epub 2007 May 21. PMID 17681163
- [Background] Hyams J, Markowitz J, Otley A, Rosh J, Mack D, Bousvaros A, Kugathasan S, Pfefferkorn M, Tolia V, Evans J, Treem W, Wyllie R, Rothbaum R, del Rosario J, Katz A, Mezoff A, Oliva-Hemker M, Lerer T, Griffiths A; Pediatric Inflammatory Bowel Disease Collaborative Research Group. Evaluation of the pediatric crohn disease activity index: a prospective multicenter experience. J Pediatr Gastroenterol Nutr. 2005 Oct;41(4):416-21. doi: 10.1097/01.mpg.0000183350.46795.42. PMID 16205508
- [Background] March JS, Parker JD, Sullivan K, Stallings P, Conners CK. The Multidimensional Anxiety Scale for Children (MASC): factor structure, reliability, and validity. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):554-65. doi: 10.1097/00004583-199704000-00019. PMID 9100431
- [Background] Walker LS, Greene JW. The functional disability inventory: measuring a neglected dimension of child health status. J Pediatr Psychol. 1991 Feb;16(1):39-58. doi: 10.1093/jpepsy/16.1.39. PMID 1826329
- [Background] Otley AR, Griffiths AM, Hale S, Kugathasan S, Pfefferkorn M, Mezoff A, Rosh J, Tolia V, Markowitz J, Mack D, Oliva-Hemker M, Wyllie R, Rothbaum R, Bousvaros A, Del Rosario JF, Evans J, Blanchard W, Hyams J; Pediatric IBD Collaborative Research Group. Health-related quality of life in the first year after a diagnosis of pediatric inflammatory bowel disease. Inflamm Bowel Dis. 2006 Aug;12(8):684-91. doi: 10.1097/00054725-200608000-00003. PMID 16917222
- [Background] Streisand R, Braniecki S, Tercyak KP, Kazak AE. Childhood illness-related parenting stress: the pediatric inventory for parents. J Pediatr Psychol. 2001 Apr-May;26(3):155-62. doi: 10.1093/jpepsy/26.3.155. PMID 11259517
- [Background] Kovacs M. The Children's Depression, Inventory (CDI). Psychopharmacol Bull. 1985;21(4):995-8. No abstract available. PMID 4089116
- [Background] Bernstein CN, Wajda A, Svenson LW, MacKenzie A, Koehoorn M, Jackson M, Fedorak R, Israel D, Blanchard JF. The epidemiology of inflammatory bowel disease in Canada: a population-based study. Am J Gastroenterol. 2006 Jul;101(7):1559-68. doi: 10.1111/j.1572-0241.2006.00603.x. PMID 16863561
- [Background] Mackner LM, Crandall WV, Szigethy EM. Psychosocial functioning in pediatric inflammatory bowel disease. Inflamm Bowel Dis. 2006 Mar;12(3):239-44. doi: 10.1097/01.MIB.0000217769.83142.c6. PMID 16534426
- [Background] Lyons, JS. Communimetrics. A communication theory of measurement for human services. New York: Springer, 2009.
- [Background] Han, C, Zhao N, Blank M, Gasink, C. Impact of psychiatric disorders on patients with crohn's disease: An analysis based on a healthcare claims database. Gastroenterology-Supplements 2010; 138(5), S-9.
- [Background] Kathol, R.G., Perez, R., Cohen, J.S., (2010). The Integrated Case Management Model: Assisting Complex Patients Regain Physical and Mental Health, Springer Publishing Co. N,Y,.
- [Background] Achenbach TM, Rescorla LA. Manual for ASEBA School-Age Forms & Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families. 2001.
- [Background] McCubbin H, Patterson J. Family Inventory of Life Events and changes. In McCubbin H, Thompson A, eds. Family assessment inventories for research and practice, pp 81-100. Madison.: University of Wisconsin, 1991.
- [Background] McCubbin H, Comeau J. Family Inventory of Resources for Management. In McCubbin H, Thompson A, eds. Family assessment inventories for research and practice, pp. 81-100. Madison: University of Wisconsin, 1991.

RESULTS

PARTICIPANT FLOW:
Groups:
- Children and Youth With IBD: Children/youth (ages 8-17) with confirmed diagnoses of Inflammatory Bowel Disease (IBD).
Period: Overall Study
Arm/Group | Children and Youth With IBD
Started | 148
Completed | 148
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Children and youth (ages of 8-17) followed in the IBD Clinic at the Children's Hospital of Eastern ONtario with confirmed diagnoses of IBD (Crohn's disease or ulcererative colitis).
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 148
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14.00 [10.25 to 17.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 89
Region of Enrollment [Number; unit: participants]
  Canada | 148

OUTCOME MEASURES:

1. Primary Outcome: Pediatric INTERMED- Complexity Index
Description: 34 item screening tool which identifies biological, psychological, social, caregiver/family and health service needs that contribute to case complexity. Each item is rated on a scale from 0-3 (0= no need to act; 1= watchful waiting or preventive intervention, 2=need for action, 3=need for immediate action).
  Minimum total score is 0 and Maximum score would be 102 (high complexity). Items on the Pediatric INTERMED are organized into 5 domains:
  Biological Domain (6 items). Minimum score is 0 and maximum score is 18 (high biological complexity).
  Psychological Domain (9 items). Minimum score is 0 and maximum score is 27 (high psychological complexity).
  Social Domain (7 items). Minimum score is 0 and maximum score is 21 (high social complexity).
  Family/Caregiver Domain (7 items). Minimum score is 0 and maximum score is 21 (high family/caregiver complexity).
  Health Services Domain (5 items). Minimum score is 0 and maximum score is 15 (high health service complexity).
Time Frame: Time of Study Participation (Completion of Pediatric INTERMED tool)
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 148
scores on a scale
  Total Complexity Index | 24 [8.25 to 39.75]
  Pediatric INTERMED Biological Domain Score | 9.0 [6 to 12]
  Pediatric INTERMED Psychological Domain Score | 4.0 [0 to 10]
  Pediatric INTERMED Social Domain Score | 4.0 [0 to 9]
  Pediatric INTERMED Caregiver/Family Domain Score | 4.0 [0 to 8.0]
  Pediatric INTERMED Health Service Domain Score | 3.0 [1.0 to 5.0]
Statistical Analysis 1: Comparison: Children and Youth With IBD; Test type: Superiority or Other; Inter-rater reliability = .87 — Inter rater reliability for a subset of 40 patients whose Pediatric INTERMED was scored by two trained raters. The median inter-rater reliability coefficient was .87
Statistical Analysis 2: Comparison: Children and Youth With IBD; Test type: Superiority or Other; Cronbach's Alpha = .91 — Overall internal consistency of the overall Pediatric INTERMED scale (34 items)

2. Primary Outcome: Correlations Between Pediatric INTERMED Domain Scores
Description: Refer to Outcome Measure 1 for information pertaining to Pediatric INTERMED domain scores.
Time Frame: Pediatric INTERMED scores at time of study participation
Measure: Number; unit: Correlation Coefficient
Groups:
- Biological: Sum of Biological Domain Item Scores
- Psychological: Sum of Psychological Domain Item Scores
- Social: Sum of Social Domain Item Scores
- Family/Caregiver: Sum of Family/Caregiver Domain Item Scores
- Health Service: Sum of Health Service Domain Item Scores
Arm/Group | Biological | Psychological | Social | Family/Caregiver | Health Service
Number analyzed (Participants) | 148 | 148 | 148 | 148 | 148
Correlation Coefficient
  Biological | 1 | .29 | .34 | .32 | .19
  Psychological | .29 | 1 | .65 | .64 | .42
  Social | .34 | .65 | 1 | .63 | .41
  Caregiver/Family | .32 | .64 | .63 | 1 | .53
  Health Service | .19 | .42 | .41 | .53 | 1
Statistical Analysis 1: Comparison: Biological vs Psychological; Test type: Superiority or Other; p < 0.05, Pearson Correlation Coefficients — Correlation between the biological and psychological domain scores on the Pediatric INTERMED. The threshold for significance is p< .05
Statistical Analysis 2: Comparison: Biological vs Social; Correlation between the Biological and Social domain scores on the Pediatric INTERMED; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 3: Comparison: Biological vs Family/Caregiver; Correlation between the Biological and Family/Caregiver Pediatric INTERMED domain scores; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 4: Comparison: Biological vs Health Service; Correlation between Biological and Health Service Pediatric INTERMED domain scores; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 5: Comparison: Psychological vs Social; Correlation between Psychology and Social Pediatric INTERMED domain scores; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 6: Comparison: Psychological vs Family/Caregiver; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 7: Comparison: Psychological vs Health Service; Correlation between Pediatric INTERMED Psychological and Health Service Pediatric INTERMED domain scores; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 8: Comparison: Social vs Family/Caregiver; Correlation between Social and Family/Caregiver Pediatric INTERMED domain scores; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 9: Comparison: Social vs Health Service; Correlation between Social and Health Service Pediatric INTERMED domain scores; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 10: Comparison: Family/Caregiver vs Health Service; Correlation between Family/Caregiver and Health Service Pediatric INTERMED domain scores; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05

3. Primary Outcome: Pediatric INTERMED Items
Description: Refer to Outcome Measure 1 for information pertaining to Pediatric INTERMED items.
Time Frame: Day 1 (At time of Pediatric Intermed Interview)
Measure: Number; unit: Percentage of participants
Groups:
- Score of 0: Rating of 0 (No Vulnerability/Need for Action) on Pediatric INTERMED Item
- Score of 1: Rating of 1 (Mild Vulnerability/Need for watchful waiting or preventive intervention) on Pediatric INTERMED item.
- Score of 2 or 3: Rating of 2 (Moderate Vulnerability/Need for Action or Development of an Intervention Plan) on the Pediatric INTERMED item or Rating of 3 (Severe Vulnerability/Need for Immediate Action of Intensive Action/Plans).
Arm/Group | Score of 0 | Score of 1 | Score of 2 or 3
Number analyzed (Participants) | 148 | 148 | 148
Percentage of participants
  Biological: Chronicity | .7 | 1.4 | 98
  Biological: Diagnostic Dilemma | .7 | 20.9 | 78.4
  Biological: Symptom Severity | 26.4 | 46.6 | 27
  Biological: Diagnostic Challenge | 60.8 | 20.9 | 18.2
  Biological: Therapeutic Complexity | 2.7 | 6.1 | 91.2
  Biological: Complications and Life Threat | 2.7 | 73.6 | 23.7
  Psychological: Barriers to Coping | 37.8 | 45.9 | 16.2
  Psychological: Resiliency | 43.9 | 43.2 | 12.8
  Psychological: Mental Health History | 51.4 | 30.4 | 18.2
  Psychological: Cogntive/Intellectual Development | 79.7 | 17.6 | 2.7
  Psychological: Adverse Developmental Events | 84.5 | 12.8 | 2.7
  Psychological: Resistance to Treatment | 49.3 | 41.9 | 8.8
  Psychological: Mental Health Symptoms | 36.5 | 53.4 | 10.2
  Psychological: Cogntive/Functinonal Impairment | 96.6 | 2.7 | .7
  Psychological: Mental Health/Cognitive Threat | 31.8 | 58.1 | 10.1
  Social: School Functionning | 36.5 | 43.9 | 19.6
  Social: Social Functioning | 63.5 | 24.3 | 12.2
  Social: Child/Youth Supports | 77.7 | 21.6 | .7
  Social: School Attendance | 55.4 | 25 | 19.6
  Social: Educational NEeds | 54.1 | 27.7 | 18.3
  Social: Community Participation | 61.5 | 28.4 | 10.2
  Social System Vulnerability | 37.8 | 52 | 10.2
  Family: Family Relationships | 58.8 | 33.1 | 8.1
  Family: Caregiver Health/Function | 45.3 | 43.9 | 10.8
  Family: Residential Stability | 60.1 | 33.8 | 6.1
  Family: Caregiver/Family Support | 61.5 | 25.7 | 12.8
  Family: Family Stress | 14.9 | 66.9 | 18.2
  Family: Parental Skills | 62.8 | 34.5 | 2.7
  Family/Caregiver System Vulnerability | 39.2 | 55.4 | 5.4
  Health System: Access to Health Care | 57.4 | 38.5 | 4.1
  Health System: Treatment Experience | 51.4 | 43.2 | 5.4
  Health System: Organization of Care | 2 | 81.1 | 16.9
  Health System: Coordination of Care | 70.9 | 25 | 4.1
  Health System Impediments | 34.5 | 61.5 | 4.1

4. Primary Outcome: IBD Disease Severity
Description: IBD Disease Severity Index categorizes patient's level of disease severity based on patient scores on the Pediatric Crohn's Disease Activity Index (PCDAI): (Hymans, Markowitz, Otley et al., 2005) and the Pediatric Ulcerative Colitis Activity Index (PUCAI) (Turner, Otley, Mack et al., 2007). Children's scores on either of these indices are used to categorize the severity of their disease as: inactive, mild, moderate, or severe.
Time Frame: Day 1 (Date of patient's participation in the Pediatric Intermed interview).
Measure: Number; unit: percentage of participants
Groups:
- Disease Severity: Remission/Inactive: Disease Severity classified as in remission/inactive
- Disease Severity: Mild: Disease Severity classified as mild
- Disease Severity: Moderate: Disease Severity classified as moderate
- Disease Severity: Severe: Disease Severity classified as severe
Arm/Group | Disease Severity: Remission/Inactive | Disease Severity: Mild | Disease Severity: Moderate | Disease Severity: Severe
Number analyzed (Participants) | 148 | 148 | 148 | 148
percentage of participants
  Disease Severity at Pediatric INTERMED Interview | 62.8 | 25.7 | 8.1 | 3.4
  Disease Severity at Diagnosis | 4.3 | 25.7 | 32.1 | 37.9

5. Primary Outcome: Time Since IBD Diagnosis
Description: Time since subject's initial IBD diagnosis. Data for each subject was obtained from chart review and was coded in "months since date of diagnosis", with a range from 1 - 131 months.
Time Frame: Data collected through chart review at time of Pediatric INTERMED interview.
Measure: Number; unit: Percentage of Participants
Groups:
- Less Than 6 Months: Less than 6 months since initial IBD diagnosis.
- 6 Months-1 Year: 6 months to 1 year since initial IBD diagnosis.
- 1 Year-5 Years: 1 - 5 years since initial IBD diagnosis.
- Greater Than 5 Years: Greater than 5 years since initial IBD diagnosis.
Arm/Group | Less Than 6 Months | 6 Months-1 Year | 1 Year-5 Years | Greater Than 5 Years
Number analyzed (Participants) | 148 | 148 | 148 | 148
Percentage of Participants | 15.5 | 34.5 | 32.4 | 17.6

6. Primary Outcome: Disease Course and Treatment
Description: Number of hospitalizations since diagnosis (total number recorded in health record), number of surgeries since diagnosis (total number recorded in health record), number of courses of Prednisone (total number recorded in health record).
Time Frame: Data collected through chart review with respect to the period since diagnosis and Day 1 (date that patient's participation in Pediatric Intermed interview)
Measure: Median (Full Range); unit: number of times it occurred
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 148
number of times it occurred
  Number of Hospitalizations since Diagnosis | 1 [0 to 11]
  Number of Surgeries Since Diagnosis | 0 [0 to 4]
  Number of Courses of Prednisone | 1 [0 to 5]

7. Primary Outcome: IBD Treatment With Immunomodulators or Anti-TNFa Medications
Description: Use of Immunomodulators (azathioprine or methotrexate). Coded for each participant as "yes" (Score of 1) or "no" (Score of 2). Use of anti-Tumor Necrosis Factor alpha (TNFa) medications (infliximab or adalimumab). Coded for each participant as "yes" (Score of 1) or "no" (Score of 2).
Time Frame: Information from review of participants chart from time of diagnosis until study participation (date of Pediatric INTERMED interview).
Measure: Number; unit: Percentage of participants treated
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 148
Percentage of participants treated
  Use of Immunomodulators | 55.4
  Use of anti-TNFa Medications | 42.6

8. Primary Outcome: Functional Disability Inventory
Description: Functional Disability Inventory: (FDI); Walker & Greene, 1991). The FDI assesses illness related activity limitations in children and adolescents. The measure consists of 15 items that are scored by the child and parent as (0) "no trouble" to "(4) "impossible". The minimum score is 0 and the maximum score is 60, with higher scores indicating greater functional disability. The FDI has demonstrated good psychometric properties with test-retest reliability of .92 and .85 at the 3-month follow-up. Concurrent validity was provided by correlation (r=.52, p<.001) between the FDI and an objective index of disability (Walker & Greene, 1991).
Time Frame: Day 1 (Date of patient's participation in the Pediatric Intermed interview).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 145
units on a scale
  FDI - Child Report | 4 [0 to 45]
  FDI- Parent Report | 2 [0 to 44]

9. Primary Outcome: Impact-III: Quality of Life Questionnaire for Children With Inflammatory Bowel Disease.
Description: 35-item self report measure for assessing quality of life in children with IBD (Otley, Griffiths, Hale et al., 2006). Items are rated on a 5-point Likert scale, with lower scores indicating poorer health related quality of life. Scores can range from 35-175. Four factor scores can be calculated: General Well-Being, Emotional Functioning, Social Functioning, Body Image, as well as a Total Quality of Life Score (Perrin, Kuhlthau, Chughtai et al., 2008).
Time Frame: Day 1 (At time of Pediatric Intermed Interview)
Population: The number of participants was lower due to some missing data for this indicator, due to a few participants not completing this questionnaire.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 142
units on a scale
  Impact III: Emotional Functioning | 45 [35.75 to 54.25]
  Impact III: Social Interactions | 22 [18 to 26]
  Impact III: General Well-Being | 57 [43.50 to 70.50]

10. Primary Outcome: Child Behaviour Checklist
Description: Child Behaviour Checklist: (CBCL: Achenbach 1991). The CBCL is used to evaluate behaviour problems and social competencies of children 6 to 18 years old. The measure is completed by parents or parent surrogates who base their ratings on the preceding 6 months. It is comprised of 120 problem items that factor into eight syndrome scales, which can be grouped into Internalizing, Externalizing and Total Problem Scales. Higher scores indicate greater level of emotional/behavioural difficulties. In the present study we utilized the following CBCL subscale scores: Internalizing, Externalizing, Social Competence, Activities Competence, Academic Competence. All scores reported are scaled to T Scores.
Time Frame: Day 1 (Date of patient's participation in the Pediatric Intermed interview).
Population: The number of participants was lower due to some missing data for this indicator, as a result of a few parents not having completed this questionnaire.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale - T Scores
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 136
Units on a Scale - T Scores
  CBCL Internalizing | 54 [39 to 69]
  CBCL Externalizing | 46 [32 to 50]
  CBCL Social Competence | 45 [34.50 to 55.50]
  CBCL Activities Competence | 48 [34 to 62]
  CBCL Academic Competence | 50 [38.5 to 51.5]

11. Primary Outcome: Children's Depression Inventory
Description: 27 item self-report questionnaire used to measure depressive symptoms in children and youth (Kovacs 1992). Each item is rated on a 3-point Likert scale (0-2) with a minimum score of 0 and a maximum score of 54, with higher scores indicating more depressive symptoms. Raw scores were scaled to T-scores to control for age and gender differences.
Time Frame: Administered at study entry
Population: The number of participants was lower due to some missing data for this outcome measure, as a result of a few participants not having completed this questionnaire.
Measure: Median (Inter-Quartile Range); unit: Units on a Scale - T Scores
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 143
Units on a Scale - T Scores | 42 [34 to 50]

12. Primary Outcome: Multidimensional Anxiety Scale for Children
Description: Multidimensional Anxiety Scale for Children: (MASC; March et a., 1997). The MASC is a pediatric self-report scale that measures symptoms of anxiety. It consists of 39 items assessing physical symptoms of anxiety, harm avoidance, social anxiety and separation/panic. Each item is answered using a four point Likert scale ranging from (0) "never true about me" to (3) "often true about me". Total scores can range from 0 to 117. The raw total score was scaled to T-Scores to control for age and sex differences.
Time Frame: Day 1 (Date of patient's participation in the Pediatric Intermed interview).
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: units on a scale- T scores
Groups:
- Children/Youth With IBD: Children/youth (ages 8-17) with confirmed diagnoses of IBD.
Arm/Group | Children/Youth With IBD
Number analyzed (Participants) | 145
units on a scale- T scores | 50.00 [36.50 to 63.50]

13. Primary Outcome: Pediatric Inventory for Parents- Difficulty Score
Description: Pediatric Inventory for parents: (PIP; Streisand et al., 2001). The PIP is a 42-item self-report measure of parenting stress associated with caring for a medically ill child. It is the only published measure of parenting stress the specifically taps the experiences and stresses that parents face when caring for a medically ill child. The Difficulty Score - indicates parents' perception of the perceived difficulty of each stressor/item. Each item is scored on a 5 point Likert scale, with total scores ranging from 42 to 210, with higher scores indicating greater "perceived difficulty".
Time Frame: Day 1 (Date of patient's participation in the Pediatric Intermed interview).
Population: The number of participants was lower due to some missing data for this outcome measure, as a result of a few parents not having completed this questionnaire.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 133
units on a scale | 82 [42.5 to 121.5]

14. Primary Outcome: Family Inventory of Life Events and Changes
Description: Family Inventory of Life Events and Changes (FILE): (McCubbin & Patterson, 1991). The FILE is a 71-item, yes/no instrument that assesses chronic and recent life stress in nine areas: intra-family strains, marital strains, pregnancy and childbearing strains, finance and business strains, work-family transitions and strains, illness and family care strains, losses, transition in and out, and family and legal violations. Family members indicate whether particular stressful events have occurred. The FILE has been found to have high reliability (Cronbach's alpha=.72), good test-retest reliability, internal consistency and evidence of construct validity. Scores can range from 0-71, with higher scores indicating greater family stress.
Time Frame: Day 1 (Date of patient's participation in the Pediatric Intermed interview).
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 139
units on a scale | 7 [0 to 14]

15. Primary Outcome: Family Inventory of Resources for Management
Description: Family Inventory of Resources for Management (FIRM): (McCubbin & Comeau 1991). The FIRM was developed to assess the family's repertoire of resources. The scale is comprised of 69 items, which are responded to using a 4-point Likert scale format (0-3). The scale has been found to have good internal reliability (r=.89, Cronbach's alpha), content and concurrent validity when used in normative sample of families with chronically ill children. The possible range for the total score is from 0-207, with higher scores indicating greater family resources for management. The Financial Well-Being subscale consists of 16 items, with potential scores ranging from 0-48, with higher scores indicating greater family financial resources.
Time Frame: Day 1 (Date of patient's participation in the Pediatric Intermed interview).
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 133
units on a scale
  Firm: Total Score | 127 [99 to 155]
  FIRM: Financial Well-being Scale | 36 [24.50 to 37.50]

16. Primary Outcome: Correlations Between Pediatric INTERMED Biological Domain Score/Items and Measures of Disease Severity, Disease Treatments and Functioning
Description: Refer to Outcome Measure 1 and Outcome Measure 3 for information pertaining to Pediatric INTERMED domains and items. Refer to Outcome Measure 4 for information pertaining to IBD Disease Severity. Refer to Outcome Measure 5 for information pertaining to Disease Treatments. Refer to Outcome Measure 8 for information pertaining to Functioning Disability Inventory. Refer to Outcome Measure 9 for information pertaining to the IMPACT III- Quality of Life Questionnaire.
Time Frame: Pediatric INTERMED and Functioning at study participation and Disease related indices since IBD Diagnosis
Measure: Number; unit: Correlation Coefficients
Groups:
- Pediatric INTERMED Biological Domain Score: Sum of all Pediatric INTERMED Biological domain item scores.
- Historical Biological Item: Chronicity: This item taps the extent and chronicity of child's physical health issues.
- Historical Biological Item: Diagnostic Dilemma: This item taps whether or not the child/youth has been seeking care for physical complaints across a substantial portion of their life and whether or not these complaints have been resolved.
- Current Biological Item: Symptom Severity: This item taps the severity/acuity of the child's current physical symptoms, and the extent to which they impact on current functioning.
- Current Biological Item: Diagnostic/Therapeutic Challenge: This item refers to the presence of physical symptoms that result in current diagnostic questions or therapeutic challenges.
- Current Biological Item: Therapeutic Complexity: This item taps whether a child's treatment for their disease is clear, unequivocal or non-invasive or requires more complex regimens which are perceived by the patient/caregivers to be time-consuming, demanding or aversive.
- Vulnerability Biological Item: Complications and Life Threat: This item taps the excepted functional impact of the present medical condition over the next 3-6 months based on the child' condition and experience with similar cases.
Arm/Group | Pediatric INTERMED Biological Domain Score | Historical Biological Item: Chronicity | Historical Biological Item: Diagnostic Dilemma | Current Biological Item: Symptom Severity | Current Biological Item: Diagnostic/Therapeutic Challenge | Current Biological Item: Therapeutic Complexity | Vulnerability Biological Item: Complications and Life Threat
Number analyzed (Participants) | 148 | 148 | 148 | 148 | 148 | 148 | 148
Correlation Coefficients
  Disease Severity at Diagnosis | -.06 | .06 | -.12 | .09 | -.15 | .04 | -.02
  Disease Severity at Study Enrolment | .36 | .01 | -.08 | .53 | .20 | .17 | .18
  Functional Disability Index- Child Rating | .50 | .16 | .00 | .56 | .20 | .03 | .23
  Functional Disability Index - Parent Rating | .52 | .27 | -.10 | .51 | .14 | .09 | .27
  Impact III: General Well-Being Scale | -.45 | -.05 | .03 | -.65 | -.24 | -.01 | -.17
  Number of Surgeries since Diagnosis | .00 | .10 | .15 | .02 | .09 | -.14 | .13
  Number of Courses of Prednisone since Diagnosis | .10 | .08 | .06 | -.01 | -.10 | .18 | -.07
  Use of Chemical Immunomodulators since Diagnosis | -.11 | -.18 | -.11 | .16 | .07 | -.42 | -.20
  Use of Biological Immunodulators Since Diagnosis | -.09 | .13 | -.04 | -.09 | .12 | -.32 | -.06
Statistical Analysis 1: Comparison: Pediatric INTERMED Biological Domain Score; Correlation between Pediatric INTERMED Biological Domain Score and IBD Disease Severity at Diagnosis; Test type: Superiority or Other; p > 0.05, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 2: Comparison: Pediatric INTERMED Biological Domain Score; Correlation between Pediatric INTERMED Biological Domain Score and IBD Disease Severity (at time of Study Participation); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 3: Comparison: Pediatric INTERMED Biological Domain Score; Correlation between Pediatric INTERMED Biological Domain Score and Functional Disability Index (child rating); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p< .05
Statistical Analysis 4: Comparison: Pediatric INTERMED Biological Domain Score; Correlation between Pediatric INTERMED Biological Domain Score and Functional Disability Index (parent rating); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<.05
Statistical Analysis 5: Comparison: Pediatric INTERMED Biological Domain Score; Correlation between Pediatric INTERMED Biological Domain Score and Impact Quality of Life: General Well Being scale; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 6: Comparison: Pediatric INTERMED Biological Domain Score; Correlation between Pediatric INTERMED Biological Domain Score and Number of Surgeries; Test type: Superiority or Other; p > 0.05, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 7: Comparison: Pediatric INTERMED Biological Domain Score; Correlation between Pediatric INTERMED Biological Domain Score and Number of Courses of Prednisone; Test type: Superiority or Other; p > 0.05, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 8: Comparison: Pediatric INTERMED Biological Domain Score; Correlation between Pediatric INTERMED Biological Domain Score and Use of Immunomodulators; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 9: Comparison: Pediatric INTERMED Biological Domain Score; Correlation between Pediatric INTERMED Biological Domain Score and Use of ant-TNFa medications; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 10: Comparison: Historical Biological Item: Chronicity; Correlation between Pediatric INTERMED Chronicity Item (Historical Biological) and Disease Severity at Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 11: Comparison: Historical Biological Item: Chronicity; Correlation between Pediatric INTERMED Chronicity Item (Historical Biological) and Disease Severity at time of study participation (Pediatric INTERMED interview); Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 12: Comparison: Historical Biological Item: Chronicity; Correlation between Pediatric INTERMED Chronicity Item (Historical Biological) and Functional Disability Index (Child Report); Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 13: Comparison: Historical Biological Item: Chronicity; Correlation between Pediatric INTERMED Chronicity Item (Historical Biological) and Functional Disability Index (Parent); Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 14: Comparison: Historical Biological Item: Chronicity; Correlation between Pediatric INTERMED Chronicity Item (Historical Biological) and Impact Quality of Life: General Well-Being; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 15: Comparison: Historical Biological Item: Chronicity; Correlation between Pediatric INTERMED Chronicity Item (Historical Biological) and Number of Surgeries; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 16: Comparison: Historical Biological Item: Chronicity; Correlation between Pediatric INTERMED Chronicity Item (Historical Biological) and Number of Courses of Prednisone; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 17: Comparison: Historical Biological Item: Chronicity; Correlation between Pediatric INTERMED Chronicity Item (Historical Biological) and Use of Immunomodulators (azathioprine or methotrexate); Test type: Superiority or Other; p < 0.05, Spearman Correlation Coefficent — The threshold for significance is p< 0.05
Statistical Analysis 18: Comparison: Historical Biological Item: Chronicity; Correlation between Pediatric INTERMED Chronicity Item (Historical Biological) and use of anti-TNFa medications; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 19: Comparison: Current Biological Item: Symptom Severity; Correlation between Pediatric INTERMED "Symptom Severity" Item (Current/Biological) and Disease Severity at Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 20: Comparison: Current Biological Item: Symptom Severity; Correlation between Pediatric INTERMED "Symptom Severity" Item (Current Biological) and IBD Disease Severity at time of study participation; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 21: Comparison: Current Biological Item: Symptom Severity; Correlation between Pediatric INTERMED "Symptom Severity" Item (Current Biological) and Functional Disability Index (child rating); Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 22: Comparison: Current Biological Item: Symptom Severity; Correlation between Pediatric INTERMED "Symptom Severity" Item (Current Biological) and Functional Disability Index (Parent Rating); Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 23: Comparison: Current Biological Item: Symptom Severity; Correlation between Pediatric INTERMED "Symptom Severity" Item (Current Biological) and Impact Quality of Life: General Well-Being Scale; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 24: Comparison: Current Biological Item: Symptom Severity; Correlation between Pediatric INTERMED "Symptom Severity" Item (Current/Biological) and Number of Surgeries; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 25: Comparison: Current Biological Item: Symptom Severity; Correlation between Pediatric INTERMED "Symptom Severity" Item (Current/Biological) and Number of Courses of Prednisone; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 26: Comparison: Current Biological Item: Symptom Severity; Correlation between Pediatric INTERMED "Symptom Severity" Item (Current/Biological) and Use of Immunomodulators; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 27: Comparison: Current Biological Item: Symptom Severity; Correlation between Pediatric INTERMED "Symptom Severity" Item (Current/Biological) and Use of anti-TNFa Medications; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 28: Comparison: Historical Biological Item: Diagnostic Dilemma; Correlations between Pediatric INTERMED "Diagnostic Dilemma" Item (Historical Biological) and Functional Disability Index (Parent) and each of the following variables: Disease Severity at Diagnosis, Disease Severity at Interview, Functional Disability Index - Child, Functional Disability Index- Parent, Impact Quality of Life: General Well Being, Number of Surgeries, Number of Courses of Prednisone, Use of Immunomodulators, Use of Anti-TNFa Medications; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05. The P-Value indicated above was found for all the correlations which were examined
Statistical Analysis 29: Comparison: Current Biological Item: Diagnostic/Therapeutic Challenge; Correlation between Pediatric INTERMED "Diagnostic/Therapeutic Challenge" Item (Current Biological) and IBD Disease Severity at Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 30: Comparison: Current Biological Item: Diagnostic/Therapeutic Challenge; Correlation between Pediatric INTERMED "Diagnostic/Therapeutic Challenge" Item (Current Biological) and IBD Disease Severity at time of study participation; Test type: Superiority or Other; p < 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 31: Comparison: Current Biological Item: Diagnostic/Therapeutic Challenge; Correlation between Pediatric INTERMED "Diagnostic/Therapeutic Challenge" Item (Current Biological) and Functional Disability Index (Child Rating); Test type: Superiority or Other; p < 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 32: Comparison: Current Biological Item: Diagnostic/Therapeutic Challenge; Correlation between Pediatric INTERMED "Diagnostic/Therapeutic Challenge" Item (Current Biological) and Functional Disability Index (parent rating); Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 33: Comparison: Current Biological Item: Diagnostic/Therapeutic Challenge; Correlation between Pediatric INTERMED "Diagnostic/Therapeutic Challenge" Item (Current Biological) and Impact Quality of LIfe: General Well-Being Scale; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 34: Comparison: Current Biological Item: Diagnostic/Therapeutic Challenge; Correlation between Pediatric INTERMED "Diagnostic/Therapeutic Challenge" Item (Current Biological) and Number of Surgeries; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 35: Comparison: Current Biological Item: Diagnostic/Therapeutic Challenge; Correlation between Pediatric INTERMED "Diagnostic/Therapeutic Challenge" Item (Current Biological) and Number of Courses of Prednisone; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 36: Comparison: Current Biological Item: Diagnostic/Therapeutic Challenge; Correlation between Pediatric INTERMED "Diagnostic/Therapeutic Challenge" Item (Current Biological) and Use of Immunomodulators; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 37: Comparison: Current Biological Item: Diagnostic/Therapeutic Challenge; Correlation between Pediatric INTERMED "Diagnostic/Therapeutic Challenge" Item (Current Biological) and Use of anti-TNFa Medications; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 38: Comparison: Current Biological Item: Therapeutic Complexity; Correlation between Pediatric INTERMED "Therapeutic Complexity" Item (Current Biological) and Disease Severity at Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 39: Comparison: Current Biological Item: Therapeutic Complexity; Correlation between Pediatric INTERMED "Therapeutic Complexity" Item (Current Biological) and Disease Severity at time of study participation (Pediatric INTERMED interview); Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 40: Comparison: Current Biological Item: Therapeutic Complexity; Correlation between Pediatric INTERMED "Therapeutic Complexity" Item (Current Biological) and Functional Disability Index (Child Rating); Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 41: Comparison: Current Biological Item: Therapeutic Complexity; Correlation between Pediatric INTERMED "Therapeutic Complexity" Item (Current Biological) and Functional Disability Index (Parent Rating); Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 42: Comparison: Current Biological Item: Therapeutic Complexity; Correlation between Pediatric INTERMED "Therapeutic Complexity" Item (Current Biological) and Impact Quality of Life: General Well-Being; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 43: Comparison: Current Biological Item: Therapeutic Complexity; Correlation between Pediatric INTERMED "Therapeutic Complexity" Item (Current Biological) and Number of Surgeries; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 44: Comparison: Current Biological Item: Therapeutic Complexity; Correlation between Pediatric INTERMED "Therapeutic Complexity" Item (Current Biological) and Number of Courses of Prednisone since diagnosis; Test type: Superiority or Other; p < 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 45: Comparison: Current Biological Item: Therapeutic Complexity; Correlation between Pediatric INTERMED "Therapeutic Complexity" Item (Current Biological) and Use of Immunomodulators (azathioprine or methotrexate); Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significiance is p<0.01
Statistical Analysis 46: Comparison: Current Biological Item: Therapeutic Complexity; Correlation between Pediatric INTERMED "Therapeutic Complexity" Item (Current Biological) and Use of ant-TNFa Medications (infliximab or adalimumab); Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The Threshold for significance is p<0.05)
Statistical Analysis 47: Comparison: Vulnerability Biological Item: Complications and Life Threat; Correlation between Pediatric INTERMED "Complications and Life Threat" Item (Vulnerability Biological) and Disease Severity at diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 48: Comparison: Vulnerability Biological Item: Complications and Life Threat; Correlation between Pediatric INTERMED "Complications and Life Threat" Item (Vulnerability Biological) and Disease Severity at study participation; Test type: Superiority or Other; p < 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 49: Comparison: Vulnerability Biological Item: Complications and Life Threat; Correlation between Pediatric INTERMED "Complications and Life Threat" Item (Vulnerability Biological) and Functional Disability Index (Child Rating); Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 50: Comparison: Vulnerability Biological Item: Complications and Life Threat; Correlation between Pediatric INTERMED "Complications and Life Threat" Item (Vulnerability Biological) and Functional Disability Index (parent rating); Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.01
Statistical Analysis 51: Comparison: Vulnerability Biological Item: Complications and Life Threat; Correlation between Pediatric INTERMED "Complications and Life Threat" Item (Vulnerability Biological) and Impact Quality of Life: General Well Being Scale; Test type: Superiority or Other; p < 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 52: Comparison: Vulnerability Biological Item: Complications and Life Threat; Correlation between Pediatric INTERMED "Complications and Life Threat" Item (Vulnerability Biological) and Number of Surgeries; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 53: Comparison: Vulnerability Biological Item: Complications and Life Threat; Correlation between Pediatric INTERMED "Complications and Life Threat" Item (Vulnerability Biological) and Number of Courses of Prednisone; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 54: Comparison: Vulnerability Biological Item: Complications and Life Threat; Correlation between Pediatric INTERMED "Complications and Life Threat" Item (Vulnerability Biological) and Use of Immunomodulators (azathioprine or methotrexate); Test type: Superiority or Other; p < 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 55: Comparison: Vulnerability Biological Item: Complications and Life Threat; Correlation between Pediatric INTERMED "Complications and Life Threat" Item (Vulnerability Biological) and Use of anti-TNFa Medications; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05

17. Primary Outcome: Correlations Between Pediatric Psychological, Social and Family Domain Scores and Measures of Emotional, Behavioural, Social and Family Functioning.
Description: Relations between Pediatric INTERMED Psychological, Social and Family Domain scores and other validated measures of subjects' psychosocial adjustment, including depression (Children's Depression Inventory- Outcome Measure 11), anxiety (Multidimensional Anxiety Scale for Children-Outcome Measure 12), Behavioural Adjustment (Internalizing and Externalizing Scores on the CBCL- Outcome Measure 10), Competence (Social, Activities and School Competence Scores from the CBCL- Outcome Measure 10), and family functioning (Parenting Inventory for Parents- Outcome Measure 13, Family Inventory of Life Events-Outcome Measure 14, Family Inventory of Resources for Management- Outcome Measure 15), and IBD health-related quality of life (IMPACT III: Emotional Functioning and Social Interactions scales- Outcome Measure 9).
Time Frame: Day 1 (Time of Study Participation)
Measure: Number; unit: Pearson Correlation Coefficient
Groups:
- Pediatric INTERMED Psychological Domain Score: Sum of Pediatric INTERMED Psychological Domain item scores
- Pediatric INTERMED Social Domain Score: Sum of Pediatric INTERMED Social Domain items scores
- Pediatric INTERMED Caregiver/Family Domain Score: Sum of Pediatric INTERMED Caregiver/Family Domain item scores
Arm/Group | Pediatric INTERMED Psychological Domain Score | Pediatric INTERMED Social Domain Score | Pediatric INTERMED Caregiver/Family Domain Score
Number analyzed (Participants) | 133 | 133 | 133
Pearson Correlation Coefficient
  CBCL Internalizing Score | .56 | .46 | .46
  CBCL Externalizing Score | .52 | .42 | .38
  Children's Depression Inventory | .41 | .46 | .38
  Multidimensional Anxiety Scale for Children | .24 | .19 | .14
  Impact III: Emotional Functioning | -.35 | -.30 | -.33
  CBCL Social Competence | -.32 | -.38 | -.29
  CBCL Activities Competence | -.18 | -.23 | -.27
  CBCL Academic Competence | -.50 | -.59 | -.35
  Impact III: Social Interactions | .40 | -.38 | -.37
  PIP Difficulty Score | .22 | .41 | .39
  Family Inventory of Life Events | .31 | .36 | .41
  Family Inventory of Resources for Management | -.26 | -.28 | -.46
Statistical Analysis 1: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Internalizing Problems (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 2: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Externalizing Problems (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 3: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Children's Depression Inventory: Total Score; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 4: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Multidimensional Anxiety Scale for Children: Total Score; Test type: Superiority or Other; p < 0.05, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 5: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Impact Quality of Life: Emotional Scale; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 6: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Social Competence Scale (Child Behaviour Checklist); Test type: Superiority or Other; p = 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 7: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Activities Competence Scale (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.05, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 8: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Academic Competence Scale (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 9: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Impact Quality of Life: Social Scale; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 10: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Pediatric Inventory for Parents: Difficulty Score (parenting stress); Test type: Superiority or Other; p < 0.05, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 11: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Family Inventory of Life Events (family stress measure); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 12: Comparison: Pediatric INTERMED Psychological Domain Score; Correlation between Pediatric INTERMED Psychological Domain Score (psychological needs) and Family Inventory of Resources for Management (family resources measure); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 13: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Internalizing Problems (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 14: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Externalizing Problems (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 15: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Children's Depression Inventory: Total Score; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 16: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Multidimensional Anxiety Scale for Children: Total Score; Test type: Superiority or Other; p < 0.05, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 17: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Impact Quality of Life: Emotional Scale; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 18: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Social Competence Scale (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 19: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Activities Competence Scale (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 20: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Academic Competence Scale (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 21: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Impact Quality of Life: Social Scale; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 22: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Pediatric Inventory for Parents: Difficulty Score (parenting stress); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 23: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Family Inventory of Life Events (family stress measure); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 24: Comparison: Pediatric INTERMED Social Domain Score; Correlation between Pediatric INTERMED Social Domain Score (social needs) and Family Inventory of Resources for Management (family resources measure); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 25: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Internalizing Problems (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 26: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Externalizing Problems (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 27: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Children's Depression Inventory: Total Score; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 28: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Multidimensional Anxiety Scale for Children: Total Score; Test type: Superiority or Other; p > 0.05, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 29: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; [analysis description as in outcome 17, analysis 5]; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 30: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Social Competence Scale (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 31: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Activities Competence Scale (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 32: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Academic Competence Scale (Child Behaviour Checklist); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance
Statistical Analysis 33: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Impact Quality of Life: Social Scale; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 34: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Pediatric Inventory for Parents: Difficulty Score (parenting stress); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 35: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; [analysis description as in outcome 17, analysis 11]; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 36: Comparison: Pediatric INTERMED Caregiver/Family Domain Score; Correlation between Pediatric INTERMED Caregiver/Family Domain Score (caregiver/family needs) and Family Inventory of Resources for Management (family resources measure); Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05

18. Primary Outcome: Likelihood of Being Identified as Having a Mental Health Need on the Pediatric INTERMED Mental/Cognitive Threat Item When Subject's Total MASC Score Falls in the Clinical Range.
Description: This outcome examined the increase in odds of a participant being identified as being rated as having a mental health need on the Pediatric INTERMED Mental Health/Cognitive Threat item when they scored in the clinical range on the Multidimensional Anxiety Scale for Children. Refer to Outcome Measure 1 for information pertaining to Pediatric INTERMED items. Refer to Outcome Measure 12 for information pertaining to the Children's Depression Inventory. Subjects were categorized into two groups based on their scores on Pediatric INTERMED Mental Health/Cognitive Threat ITEM: low psychological need (rating of 0 or 1) and high psychological need (rating of 2 or 3). Children with T scores above 65 on the Multidimensional Anxiety Scale for Children were categorized as falling into the clinical range.
Time Frame: Day 1 (At time of Pediatric Intermed Interview)
Population: The number of participants was lower due to some missing data for the MASC measure, due to fewer participants completing this questionnaire.
Measure: Number; unit: participants
Groups:
- Subjects With MASC Scores in the Clinical Range.: Children whose scores on the Multidimensional Anxiety Scale for Children fell within the clinical range.
- Subjects With MASC Scores in the Non-clinical Range: Children whose scores on the Multidimensional Anxiety Scale for Children fell below the clinical range.
Arm/Group | Subjects With MASC Scores in the Clinical Range. | Subjects With MASC Scores in the Non-clinical Range
Number analyzed (Participants) | 145 | 145
participants
  Mental Health/Cognitive Vulnerability Need | 4 | 10
  No Mental Health/Cognitive Vulnerability | 6 | 125
Statistical Analysis 1: Comparison: Subjects With MASC Scores in the Clinical Range. vs Subjects With MASC Scores in the Non-clinical Range; Test type: Superiority or Other; Odds Ratio (OR) = 8.33, 95% CI 2-sided [2.02 to 34.47]

19. Primary Outcome: Likelihood of Being Identified as Having a Mental Health Need on the Pediatric INTERMED Mental/Cognitive Threat Item When Subject's Total Children's Depression Inventory (CDI) Score is in the Clinical Range.
Description: This outcome examined the increase in odds of a participant being identified as being rated as having a mental health need on the Pediatric INTERMED Mental Health/Cognitive Threat Item when they scored in the clinical range on the Children's Depression Inventory. Refer to Outcome Measure 1 for information pertaining to Pediatric INTERMED items. Refer to Outcome Measure 11 for information pertaining to the Children's Depression Inventory. Subjects were categorized into two groups based on their scores on Pediatric INTERMED Mental Health/Cognitive Threat ITEM: low psychological need (rating of 0 or 1) and high psychological need (rating of 2 or 3). Children with T scores above 65 on the Children's Depression Inventory were categorized as falling into the clinical range.
Time Frame: Day 1 (At time of Pediatric Intermed Interview)
Population: The number of participants was lower due to some missing data for the CDI measure, due to fewer participants completing this questionnaire.
Measure: Number; unit: participants
Groups:
- Subjects With CDI Scores in the Clinical Range.: Children whose scores on the Children's Depression Inventory fell within the clinical range.
- Subjects With CDI Scores in the Non-clinical Range: Children whose scores on the Children's Depression Inventory fell below the clinical range.
Arm/Group | Subjects With CDI Scores in the Clinical Range. | Subjects With CDI Scores in the Non-clinical Range
Number analyzed (Participants) | 143 | 143
participants
  Mental Health/Cognitive Vulnerability Need | 3 | 11
  No Mental Health/Cognitive Vulnerability | 4 | 125
Statistical Analysis 1: Comparison: Subjects With CDI Scores in the Clinical Range. vs Subjects With CDI Scores in the Non-clinical Range; Test type: Superiority or Other; Odds Ratio (OR) = 8.52, 95% CI 2-sided [1.70 to 43.02]

20. Primary Outcome: Likelihood of Being Identified as Having a Mental Health Need on the Pediatric INTERMED Mental/Cognitive Threat Item When Subject's CBCL Internalizing Score Falls in the Clinical Range.
Description: This outcome examined the increase in odds of a participant being identified as being rated as having a mental health need on the Pediatric INTERMED Mental Health/Cognitive Threat Item when they scored in the clinical range on the Child Behavior Checklist - Internalizing Problems Scale. Refer to Outcome Measure 1 for information pertaining to Pediatric INTERMED items. Refer to Outcome Measure 10 for information pertaining to the Child Behavior Checklist. Subjects were categorized into two groups based on their scores on Pediatric INTERMED Mental Health/Cognitive Threat ITEM: low psychological need (rating of 0 or 1) and high psychological need (rating of 2 or 3). Children with T scores above 63 on the Child Behavior Checklist Internalizing Scale were categorized as falling into the clinical range.
Time Frame: Day 1 (At time of Pediatric Intermed Interview)
Population: The number of participants was lower due to some missing data for the CBCL measure, due to fewer participants completing this questionnaire.
Measure: Number; unit: participants
Groups:
- CBCL Internalizing Score in the Clinical Range.: Children whose scores on the CBCL Internalizing Scale fell within the clinical range.
- CBCL Internalizing Score in the Non-clinical Range: Children's whose scores on the CBCL Internalizing Scale fell below the clinical range.
Arm/Group | CBCL Internalizing Score in the Clinical Range. | CBCL Internalizing Score in the Non-clinical Range
Number analyzed (Participants) | 135 | 135
participants
  Mental Health/Cognitive Vulnerability Need | 8 | 5
  No Mental Health/Cognitive Vulnerability | 22 | 100
Statistical Analysis 1: Comparison: CBCL Internalizing Score in the Clinical Range. vs CBCL Internalizing Score in the Non-clinical Range; Test type: Superiority or Other; Odds Ratio (OR) = 7.27, 95% CI 2-sided [2.17 to 24.36]

21. Primary Outcome: Likelihood of Being Identified as Having a Mental Health Need on the Pediatric INTERMED Mental/Cognitive Threat Item When Subject's CBCL Externalizing Score is in the Clinical Range.
Description: This outcome examined the increase in odds of a participant being identified as being rated as having a mental health need on the Pediatric INTERMED Mental Health/Cognitive Threat Item when they scored in the clinical range on the Child Behavior Checklist - Externalizing Problems Scale. Refer to Outcome Measure 1 for information pertaining to Pediatric INTERMED items. Refer to Outcome Measure 10 for information pertaining to the Child Behavior Checklist. Subjects were categorized into two groups based on their scores on Pediatric INTERMED Mental Health/Cognitive Threat ITEM: low psychological need (rating of 0 or 1) and high psychological need (rating of 2 or 3). Children with T scores above 63 on the Child Behavior Checklist Externalizing Scale were categorized as falling into the clinical range.
Time Frame: Day 1 (At time of Pediatric Intermed Interview)
Population: as for outcome 20
Measure: Number; unit: participants
Groups:
- CBCL Externalizing Score in the Clinical Range.: Children whose scores on the CBCL Externalizing scale fell within the clinical range.
- CBCL Externalizing Score in the Non-clinical Range: Children whose scores on the CBCL Externalizing Scale fell below the clinical range.
Arm/Group | CBCL Externalizing Score in the Clinical Range. | CBCL Externalizing Score in the Non-clinical Range
Number analyzed (Participants) | 135 | 135
participants
  Mental Health/Cognitive Vulnerability Need | 5 | 8
  No Mental Health/Cognitive Vulnerability | 3 | 119
Statistical Analysis 1: Comparison: CBCL Externalizing Score in the Clinical Range. vs CBCL Externalizing Score in the Non-clinical Range; Test type: Superiority or Other; Odds Ratio (OR) = 24.79, 95% CI 2-sided [5.00 to 122.84]

22. Primary Outcome: Correlations Between Pediatric Health System Domain Score/Items and Disease and Health Service Indicators
Description: Refer to Outcome Measure 1 and Outcome Measure 3 for information pertaining to Pediatric INTERMED domain scores and items. Refer to Outcome Measure 6 for information pertaining to Disease/Treatment Indicators. Refer to Outcome Measure 23 for information about the Number of Services involved in Child's Care, and to Outcome Measure 15 for information about the Family Inventory of Resources for Management.
Time Frame: Pediatric INTERMED and FIRM scores obtained at Study Entry and Disease and Health Care Indicators since IBD Diagnosis
Measure: Number; unit: Correlation Coefficients
Groups:
- Pediatric Intermed: Health System Domain Score: Sum of Pediatric INTERMED health system item scores.
- Historical Health System Item: Access to Health Care: This item refers to anything in the past that served as an obstacle, hindering the patient's access to healthcare.
- Historical Health System Item: Treatment Experience: This item describes the degree to which the child and family's prior health care experiences have been positive in terms of good outcomes and relationships with health care providers.
- Current Health System Item: Organization of Care: This item describes the nature and organization of the health care services that the child is current receiving.
- Current Health System Item: Coordination of Care: This item describes the extent to which the different health care providers working with the child are in contact with each other.
- Vulnerability Health System Item: Health System Impediments: This item anticipates the problems that the child/youth may encounter in the next 3-6 months in receiving the services he/she requires.
Arm/Group | Pediatric Intermed: Health System Domain Score | Historical Health System Item: Access to Health Care | Historical Health System Item: Treatment Experience | Current Health System Item: Organization of Care | Current Health System Item: Coordination of Care | Vulnerability Health System Item: Health System Impediments
Number analyzed (Participants) | 148 | 148 | 148 | 148 | 148 | 148
Correlation Coefficients
  Number of Services involved in Child's Care | .26 | .08 | .25 | .37 | .20 | .15
  Number of Hospitalizations since Diagnosis | .34 | .36 | .14 | .11 | .09 | .23
  Numbers of Surgeries since Hospitalization | .22 | .25 | .10 | .08 | .13 | .11
  FIRM: Financial Well Being Scale | -.32 | -.34 | -.13 | -.03 | -.15 | -.36
Statistical Analysis 1: Comparison: Pediatric Intermed: Health System Domain Score; Correlation between Pediatric INTERMED Health System Domain Score (health system needs/complexity) and Number of Hospital Services involved in the child's care; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 2: Comparison: Pediatric Intermed: Health System Domain Score; Correlation between Pediatric INTERMED Health System Domain Score (health system needs/complexity) and Number of Inpatient Hospitalizations since IBD diagnosis; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 3: Comparison: Pediatric Intermed: Health System Domain Score; Correlation between Pediatric INTERMED Health System Domain Score (health system needs/complexity) and Number of Surgeries since IBD diagnosis; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 4: Comparison: Pediatric Intermed: Health System Domain Score; Correlation between Pediatric INTERMED Health System Domain Score (health system needs/complexity) and Family Financial Well Being; Test type: Superiority or Other; p < 0.01, Pearson Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 5: Comparison: Historical Health System Item: Access to Health Care; Correlation between Pediatric INTERMED "Access to Health Care" Item (historical/health system) and Number of Hospital Services Involved in the Child's Care; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 6: Comparison: Historical Health System Item: Access to Health Care; Correlation between Pediatric INTERMED "Access to Health Care" Item (historical/health system) and Number of Hospitalizations since Child's IBD Diagnosis; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 7: Comparison: Historical Health System Item: Access to Health Care; Correlation between Pediatric INTERMED "Access to Health Care" Item (historical/health system) and Number of Surgeries since Diagnosis; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 8: Comparison: Historical Health System Item: Access to Health Care; Correlation between Pediatric INTERMED "Access to Health Care" Item (historical/health system) and Family Financial Well-Being; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 9: Comparison: Historical Health System Item: Treatment Experience; Correlation between Pediatric INTERMED "Treatment Experience" Item (historical/health system) and Number of Hospital Services Involved in the Child's Care; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 10: Comparison: Historical Health System Item: Treatment Experience; Correlation between Pediatric INTERMED "Treatment Experience" Item (historical/health system) and Number of Hospitalizations since Child's IBD Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 11: Comparison: Historical Health System Item: Treatment Experience; Correlation between Pediatric INTERMED "Treatment Experience" Item (historical/health system) and Number of Surgeries since child's diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 12: Comparison: Historical Health System Item: Treatment Experience; Correlation between Pediatric INTERMED "Treatment Experience" Item (historical/health system) and Family Financial Well-Being; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 13: Comparison: Current Health System Item: Organization of Care; Correlation between Pediatric INTERMED "Organization of Care" Item (current/health system) and Number of Hospital Services Involved in the Child's Care; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 14: Comparison: Current Health System Item: Organization of Care; Correlation between Pediatric INTERMED "Organization of Care" Item (current/health system) and Number of Hospitalizations since IBD Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 15: Comparison: Current Health System Item: Organization of Care; Correlation between Pediatric INTERMED "Organization of Care" Item (current/health system) and Number of Surgeries since Child's IBD Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 16: Comparison: Current Health System Item: Organization of Care; Correlation between Pediatric INTERMED "Organization of Care" Item (current/health system) and Family Financial Well-Being; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 17: Comparison: Current Health System Item: Coordination of Care; Correlation between Pediatric INTERMED "Coordination of Care" Item (current/health system) and Number of Hospital Services Involved in the Child's Care; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 18: Comparison: Current Health System Item: Coordination of Care; Correlation between Pediatric INTERMED "Coordination of Care" Item (current/health system) and Number of Hospitalizations since Child's IBD Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 19: Comparison: Current Health System Item: Coordination of Care; Correlation between Pediatric INTERMED "Coordination of Care" Item (current/health system) and Number of Surgeries Child's IBD Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 20: Comparison: Current Health System Item: Coordination of Care; Correlation between Pediatric INTERMED "Coordination of Care" Item (current/health system) and Family Financial Well Being; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 21: Comparison: Vulnerability Health System Item: Health System Impediments; Correlation between Pediatric INTERMED "Health System Impediments" Item (vulnerability/health system) and Number of Hospital Services Involved in the Child's Care; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 22: Comparison: Vulnerability Health System Item: Health System Impediments; Correlation between Pediatric INTERMED "Health System Impediments" Item (vulnerability/health system) and Number of Hospitalizations since Child's IBD Diagnosis. Services Involved in the Child's Care; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 23: Comparison: Vulnerability Health System Item: Health System Impediments; Correlation between Pediatric INTERMED "Health System Impediments" Item (vulnerability/health system) and Number of Surgeries since Child's IBD Diagnosis; Test type: Superiority or Other; p > 0.05, Spearman Correlation Coefficient — The threshold for significance is p<0.05
Statistical Analysis 24: Comparison: Vulnerability Health System Item: Health System Impediments; Correlation between Pediatric INTERMED "Health System Impediments" Item (vulnerability/health system) and Family Financial Well-Being; Test type: Superiority or Other; p < 0.01, Spearman Correlation Coefficient — The threshold for significance is p<0.05

23. Primary Outcome: Total Number of Hospital Services Involved in Child's Care.
Description: Measure of number of hospital services involved in each child's care during the three month period prior to the Pediatric INTERMED interview.
Time Frame: Data collected through chart review with respect to the three month period prior to Day 1 (date of patient's participation in Pediatric Intermed interview)
Measure: Median (Full Range); unit: R Square change statistic
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 148
R Square change statistic | 2.00 [0 to 5.00]
Statistical Analysis 1: Comparison: Children and Youth With IBD; A hierarchical multiple (linear) regression analysis was conducted to determine the predictive relation between the Pediatric INTERMED indicator of case complexity and the number of hospital services involved in child's care. Gender, and time since diagnosis were entered as covariates (Step 1), followed by current disease severity (Step 2) and the Pediatric INTERMED Complexity Index (Step 3). Diagnostic tests for collinearity were conducted and all assumptions for the analysis were met; Test type: Superiority or Other; p < 0.01, Regression, Linear — p<0.05 Threshold for statistical significance; Rsquare change statistic = 0.08

24. Primary Outcome: Number of Calls to IBD Nurse
Description: Total number of calls made by patient or parent to the IBD clinic nurse during the 3-month period prior to the Pediatric Intermed Interview
Time Frame: as for outcome 23
Measure: Median (Full Range); unit: Number of calls
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 148
Number of calls | 0 [0 to 15]
Statistical Analysis 1: Comparison: Children and Youth With IBD; A hierarchical multiple (linear) regression analysis was conducted to determine the predictive relation between the Pediatric INTERMED indicator of case complexity and the number of calls to the IBD Nurse. Gender, and time since diagnosis were entered as covariates (Step 1), followed by current disease severity (Step 2) and the Pediatric INTERMED Complexity Index (Step 3). Diagnostic tests for collinearity were conducted and all assumptions for the analysis were met; Test type: Superiority or Other; p < 0.01, Regression, Linear — Threshold for statistical significance is p<0.01; R2Change = .05

25. Primary Outcome: Number of Extra Appointments With the IBD Team
Description: Number of extra appointments (unscheduled, emergency) with the IBD Team during the 3 month period prior to the Pediatric INTERMED interview.
Time Frame: as for outcome 23
Measure: Median (Full Range); unit: Number of appointments
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 148
Number of appointments | 0 [0 to 4]
Statistical Analysis 1: Comparison: Children and Youth With IBD; A hierarchical multiple (linear) regression analysis was conducted to determine the predictive relation between the Pediatric INTERMED indicator of case complexity and the number of extra appointments with the IBD team. Gender, and time since diagnosis were entered as covariates (Step 1), followed by current disease severity (Step 2) and the Pediatric INTERMED Complexity Index (Step 3); Test type: Superiority or Other; p < 0.01, Regression, Linear — p<.05 threshold for statistical significance; Diagnostic tests for collinearity were conducted and all assumptions for the analysis were met; Rsquare change statistic = .05

26. Primary Outcome: Number of Visits to the Hospital Emergency Department
Description: Number of times that the patient visited the hospital Emergency Department in the 3-month period prior to the Pediatric INTERMED interview.
Time Frame: as for outcome 23
Measure: Median (Full Range); unit: Emergency Department Visits
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 148
Emergency Department Visits | 0 [0 to 5]
Statistical Analysis 1: Comparison: Children and Youth With IBD; A hierarchical multiple (linear) regression analysis was conducted to determine the predictive relation between the Pediatric INTERMED indicator of case complexity and the number of ER Visits. Gender, and time since diagnosis were entered as covariates (Step 1), followed by current disease severity (Step 2) and the Pediatric INTERMED Complexity Index (Step 3). Diagnostic tests for collinearity were conducted and all assumptions for the analysis were met; Test type: Superiority or Other; p < 0.05, Regression, Linear — Threshold for statistical significance is p <0.05; R2Change = .03

27. Primary Outcome: Number of Inpatient Hospital Admissions
Description: Total number of times that the patient was admitted to hospital during the 3-month period prior to the Pediatric INTERMED Interview.
Time Frame: as for outcome 23
Measure: Median (Full Range); unit: Number of hospital admissions
Arm/Group | Children and Youth With IBD
Number analyzed (Participants) | 148
Number of hospital admissions | 0 [0 to 3.00]
Statistical Analysis 1: Comparison: Children and Youth With IBD; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p < 0.01, Regression, Linear; R2Change = .07

ADVERSE EVENTS:
Time Frame: At time of study participation and for 6 months following this.
Arm/Group | Children and Youth With IBD
Serious Adverse Events (participants affected / at risk) | 0/148
Other Adverse Events (participants affected / at risk) | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No